CLINICAL TRIAL: NCT00081237
Title: A Phase I Study of OSI-7904L In Combination With Oxaliplatin In Patients With Advanced Colo-Rectal Cancer
Brief Title: OSI-7904L and Oxaliplatin in Treating Patients With Refractory or Recurrent Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16033; EORTC-16033; OSI-EORTC-16033
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — ((S)-2-(5-(1,2-dihydro-3-methyl-1-oxobenzo(f)-quinazoline-9-yl)methyl)amino-1-oxo-2-isoindolynyl)-glutaric acid; Oxaliplatin

INTERVENTIONS:
Drug: OSI-7904L
Drug: oxaliplatin

SUMMARY:
RATIONALE: OSI-7904L may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining OSI-7904L with oxaliplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of OSI-7904L and oxaliplatin in treating patients with refractory or recurrent advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity of OSI-7904L and oxaliplatin in patients with refractory or recurrent advanced colorectal cancer.
* Determine the maximum tolerated dose of this regimen in these patients.
* Determine a safe dose for this regimen in these patients.

Secondary

* Determine the pharmacokinetic profile of this regimen in these patients.
* Determine the safety profile of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a nonrandomized, multicenter, open-label, dose-escalation study.

Patients receive oxaliplatin IV over 2 hours followed by OSI-7904L IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of OSI-7904L and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. A maximum of 12 patients receive treatment at the MTD.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 3-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Radiologic evidence of advanced disease
* At least 1 measurable lesion at least 20 mm OR at least 10 mm by spiral CT scan

  * Indicator lesions in a previously irradiated field are allowed provided the irradiated lesion has clearly progressed OR a new lesion has developed in the irradiated field
* Failed 1, and only 1, line of prior chemotherapy for advanced/metastatic disease

  * Disease progression during chemotherapy OR within 6 months after completion of treatment
* No symptomatic brain metastases meeting any of the following criteria:

  * Unstable
  * Inadequately controlled with fixed-dose oral steroids
  * Potentially life-threatening
  * Required radiotherapy with the past 28 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* AST and ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin < 1.5 times ULN
* No hepatitis
* No cirrhosis

Renal

* Creatinine < 1.5 times ULN

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* HIV negative
* No preexisting neuropathy ≥ grade 2
* No active or uncontrolled infection
* No other serious illness or medical condition
* No chronic alcohol abuse
* No known hypersensitivity to systemic liposomal formulations or compounds chemically related to OSI-7904L or oxaliplatin
* No prior psychiatric or neurologic condition that would preclude study compliance or giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 21 days since prior immunotherapy
* At least 21 days since prior monoclonal antibody therapy

Chemotherapy

* See Disease Characteristics
* At least 21 days since prior chemotherapy and recovered*
* No prior oxaliplatin NOTE: *Alopecia allowed

Endocrine therapy

* See Disease Characteristics
* At least 21 days since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 21 days since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of bone marrow reserve

Surgery

* Recovered from prior surgery

Other

* At least 21 days since prior tyrosine kinase inhibitor therapy
* More than 21 days since prior investigational agents
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended dose for future trials as measured by CTC v3.0

SECONDARY OUTCOMES:
Safety profile as measured by CTC v3.0
Response as measured by RECIST every 6 weeks (2 courses)
Pharmacodynamics as measured by drug concentration in the blood during course 1
Time to progression as measured by Kaplan Meier and RECIST every 6 weeks during treatment and then every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoffski, MD, MPH, Study Chair — Hannover Medical School
Locations (2):
- Medizinische Hochschule Hannover, Hanover, Germany
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom

REFERENCES:
- [Result] Clamp AR, Schoffski P, Valle JW, Wilson RH, Marreaud S, Govaerts AS, Debois M, Lacombe D, Twelves C, Chick J, Jayson GC; EORTC New Drug Development Group. A phase I and pharmacokinetic study of OSI-7904L, a liposomal thymidylate synthase inhibitor in combination with oxaliplatin in patients with advanced colorectal cancer. Cancer Chemother Pharmacol. 2008 Apr;61(4):579-85. doi: 10.1007/s00280-007-0509-5. Epub 2007 May 23. PMID 17520255